CLINICAL TRIAL: NCT05680129
Title: A Phase 3, Multi-center, Open-label, Randomized Study to Evaluate the Efficacy and Safety of XW003 Versus Dulaglutide in Patients With T2DM Inadequately Controlled by Metformin
Brief Title: A Phase 3 Study to Evaluate the Efficacy of XW003 Compared With Dulaglutide in Participants With T2DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCW0502-1032
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2023-07

CONDITIONS: T2DM; Type 2 Diabetes Mellitus
Keywords: T2DM; Glucagon-like peptide-1; GLP-1; Ecnoglutide; XW003
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- B1: XW003+MET (Experimental): High dosage of XW003 once weekly
  Interventions: Drug: Ecnoglutide high dosage; Drug: Metformin
- B2: XW003+MET (Experimental): Low dosage of XW003 once weekly
  Interventions: Drug: Ecnoglutide low dosage; Drug: Metformin
- B3: Dulaglutide+MET (Active Comparator): 1.5mg Dulaglutide once weekly
  Interventions: Drug: Dulaglutide; Drug: Metformin

INTERVENTIONS:
Drug: Ecnoglutide high dosage — Administered subcutaneously
  Other Names: XW003
  Arms: B1: XW003+MET
Drug: Ecnoglutide low dosage — Administered subcutaneously
  Other Names: XW003
  Arms: B2: XW003+MET
Drug: Dulaglutide — Administered subcutaneously
  Arms: B3: Dulaglutide+MET
Drug: Metformin — Administered orally

SUMMARY:
The aim of the study is to compare the efficacy and safety of two XW003 doses versus dulaglutide as add-on therapy to metformin in participants with type 2 diabetes mellitus (T2DM)

DETAILED DESCRIPTION:
In this Phase 3 study, eligible participants will be randomized in a 1:1:1 ratio to receive once-weekly subcutaneous XW003 (high or dose) or active comparator dulaglutide as add-on to metformin treatment for 52 weeks, including a dose-escalation period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to participate in the study, give written informed consent, and comply with the study specific requirements and all protocol procedures
2. Sex: male or female; Age: 18 to 75 years, inclusive
3. BMI: 20.0 kg/m^2 to 35.0 kg/m^2, inclusive
4. Have been diagnosed with T2DM for at least 3 months and treated with a stable dose of metformin (≥1500 mg/day) in addition to diet and exercise during the 8 weeks prior to screening.
5. HbA1c ranging from 7.5% to 11.0% at screening, inclusive
6. FPG ≤13.9 mmol/L at screening

Exclusion Criteria:

1. History of type 1 or other types of diabetes mellitus
2. Use of insulin during the 6 months preceding screening
3. History of proliferative diabetic retinopathy, diabetic maculopathy, diabetic neuropathy, or diabetic foot during the 6 months prior to screening.
4. History of acute or chronic pancreatitis or high-risk factors for pancreatitis
5. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
6. History of stomach surgeries or disorders associated with slowed emptying of the stomach during the past 6 months.
7. History of heart attack, stroke or congestive heart failure of Grade 3 or 4 in the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, week 32

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Baseline, Week 5, Week 9, Week 13, Week 17, Week 25, Week 43 and Week 52
Change from baseline in fasting plasma glucose (FPG) | Baseline, Week 32 and Week 52
Change from baseline in lipid panel | Baseline, Week 32 and Week 52
Change from baseline in body weight | Baseline, Week 32 and Week 52
Pharmacokinetics: plasma trough level of XW003 | Baseline, Day 29, Day 57, Day 85, Day 224, Day 364 and Day 399

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Dr, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- ZHONGSHAN Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He Y, Mi N, Cheng Z, Xue H, Han J, Wang H, Wang H, Wu J, Shi X, Zhao S, Duan B, Zhu Y, Zhou Y, Li F, Wang X, Ling H, Wang S, Li Q, Jiang F, Yang M, Bing S, Zheng Q, Ning J, Guo M, Bu Y, Guan L, Li Y, Yang L, Guo W, Pan H, Li X. Efficacy and safety of cAMP-biased GLP-1 receptor agonist ecnoglutide versus dulaglutide in patients with type 2 diabetes and elevated glucose concentrations on metformin monotherapy (EECOH-2): a 52-week, multicentre, open-label, non-inferiority, randomised, phase 3 trial. Lancet Diabetes Endocrinol. 2025 Oct;13(10):863-873. doi: 10.1016/S2213-8587(25)00196-2. Epub 2025 Aug 22. PMID 40854315